CLINICAL TRIAL: NCT03827759
Title: Multicenter, Diagnostic and Prospective Study to Differentiate Child Septic and Inflammatory Arthritis by Comparative Analysis
Brief Title: Differentiate Children Septic and Inflammatory Arthritis by Comparative Analysis
Acronym: DIANE
Status: Terminated | Type: Observational
Why Stopped: End of the inclusion period and difficulty in recruiting the youngest patients
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0293; 7683 (Other: UH Montpellier)
Record Dates: First submitted 2019-01-23; First posted 2019-02-01 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Septic Arthritis; Inflammatory Arthritis; Children
Keywords: idiopathic juvenile arthritis, septic arthritis, biomarkers
MeSH Terms: conditions — Arthritis, Infectious; Arthritis; Arthritis, Juvenile

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Synovial liquid and blood samples (with : proteomic, MiRNA searching, multiplex cytokine analysis and cellular phenotyping) will be analysed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- septic arthritis (group A): Patients with acute juvenile arthritis with suspicion of bacterial infection,confirmed on a bacteriological plan, either by culture of the articular liquid or by blood culture, or by molecular biology in the articular liquid;
- inflammatory arthritis (group B): Patients with idiopathic juvenile arthritis
- control (group C): Healthy children who are matched by the age and at the sex in the groups A and B, to analyze elements studied in the blood.

SUMMARY:
The purpose is to found new biomarker that differentiate septic arthritis and Juvenile Idiopathic Arthritis in children. Synovial liquid and blood samples with proteomic, MiRNA searching, multiplex cytokine analysis and cellular phenotyping, will be analysed. The results for each data will be compared in function of the disease to search discriminant markers. On behalf with this result specific pathways could be identified .

DETAILED DESCRIPTION:
This a multicentric prospective study that compares biological fluids as synovial liquid and blood samples to find biomarkers that could distinguish septic arthritis and juvenile idiopathic arthritis. Prospectively, patients will be recruited under the age of 15 who are in care for septic or inflammatory arthritis at the University Hospitals of Montpellier, Lyon, Nimes and Toulouse. Patients should have an indication of blood and synovial as part of their management :

Group A: acute juvenile arthritis with suspicion of bacterial infection, , confirmed on a bacteriological plan, either by culture of the articular liquid or by blood culture, or by molecular biology in the articular liquid.

Group B: Idiopathic juvenile arthritis and control topics (Group C). In this project, the aim is to analyze all in all 50 articular liquids and serum of inflammatory arthritises (Group B), and 30 articular liquids and serum of infectious confirmed arthritises (Group A) which will require the inclusion about 50 possibly septic arthritis. The diagnosis of infectious arthritis is not immediate, he(it) is confirmed at the latest three weeks after the draining. So a group of control will be constituted.

Group C: the blood of 20 healthy children matched by the age and at the sex in the groups A and B will be collected to analyze elements studied in the blood.

* Inclusion criteria :

Group A and group B:

* Subject of more than 6 months and under age 15 years,
* Presenting acute arthritis taken care in the University Hospitals of Montpellier, Nimes, Toulouse or Lyon, and requiring an articular puncture
* Child benefiting from a social security system,
* Collection of the consent of the legal parents/representatives,

Group C:

* Subject of more than 6 months and under age 15 include
* Taken care in the University Hospital of Montpellier, and requiring a venous draining,
* Child benefiting from a social security system,
* Collection of the consent of the legal parents/representatives

  * Non inclusion criteria /

Group A and group B:

* Contraindication in an articular draining: platelet 50 000/mm3, pathologic hemostasis
* Treatment by biological therapy, corticoids or other immunosuppressant treatment in the month preceding the articular draining,
* antibiotic begun more than 24 hours before the inclusion.

Group C: ·

* Patient achieves of an inflammatory chronic pathology
* Patient having presented an infectious episode in the previous 8 days -Patients under immunosuppressor or anti-infective

Methods of measure of assessment criteria

Analysis will be done on blood samples and synovial liquid, that remains after sample collected for the management of their disease. The blood test and an synovial liquid draining will be realized at the subject. Before freezing, aliquots will be realized so that every analysis can benefit from a minimum volume:

* Cellular analyses: will be only made in Montpellier and established by the set of collected cells (no necessary volume).
* Proteomic, MiRNA analysis and cytokine dosing will been done in the second time.

Statistical analysis will be done to individualize biomarkers.

ELIGIBILITY:
Inclusion Criteria:

Group A and group B:

* Subject of more than 6 months and under age 15 years,
* Presenting acute arthritis taken care in the University Hospitals of Montpellier, Nimes, Toulouse or Lyon, and requiring an articular puncture,
* Child benefiting from a social security system,
* Collection of the consent of the legal parents/representatives,

Group C:

* Subject of more than 6 months and under age 15 include,
* Taken care in the University Hospital of Montpellier, and requiring a venous draining,
* Child benefiting from a social security system,
* Collection of the consent of the legal parents/representatives

Exclusion Criteria:

Group A and group B:

* Contraindication in an articular draining: platelet 50 000/mm3, pathologic hemostasis
* Treatment by biological therapy, corticoids or other immunosuppressant treatment in the month preceding the articular draining,
* antibiotic begun more than 24 hours before the inclusion.

Group C:

* Patient achieves of an inflammatory chronic pathology
* Patient having presented an infectious episode in the previous 8 days
* Patients under immunosuppressor or anti-infective

Ages: 6 Months to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Subjects of more than 6 months and under age 15 years, presenting acute arthritis, and control subjects
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2021-06-06 (Actual); Study Completion 2022-07-29 (Actual)

PRIMARY OUTCOMES:
Qualitative analysis of new biological markers (proteic) that discriminate inflammatory and infectious arthritis | 1 day
  Identify blood sampling proteic markers of Arthritis childhood
Qualitative analysis of new biological markers (cytokine) that discriminate inflammatory and infectious arthritis | 1 day
  Identify blood sampling markers (cytokine : interleukin 2, interleukin 4, interleukin 6, interleukin 7, tumor necrosis factor alpha (TNF)) of Arthritis childhood
Qualitative analysis of new cellular markers that discriminate inflammatory and infectious arthritis | 1 day
  Identify blood sampling cellular markers (lymphocytes and monocytes) of Arthritis childhood

SECONDARY OUTCOMES:
Qualitative analysis of inflammatory process markers | 1 day
  Identify articular liquid sampling biomarkers (lymphocytes and interleukins) of Arthritis childhood

CONTACTS AND LOCATIONS:
Overall Officials: Eric JEZIORSKI, MD PhD, Study Director — University Hospital, Montpellier
Locations (5):
- France (5):
  - CHU Montpellier - Pediatric emergencies, Montpellier, Hérault
  - Hospices Civils de Lyon - pediatric rheumatology, Lyon
  - Hôpital Saint Joseph, Marseille
  - CHU Nîmes - Pediatrics, Nîmes
  - CHU Toulouse - Pediatric infectious diseases, Toulouse